CLINICAL TRIAL: NCT02925936
Title: Choice of Tube Extremity in Emission of Lowest Radiation Dose in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Guilherme Oberto Rodrigues, Master of Science, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4769/12
Record Dates: First submitted 2016-05-12; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Radiation Absorption; Radiography
Keywords: Radiography; Radiation; Diagnostic imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cathode (Active Comparator): Thyroid facing the cathode end of xray machine
  Interventions: Other: Thyroid facing the cathode end of xray machine
- Anode (Active Comparator): Thyroid facing the anode end of xray machine
  Interventions: Other: Thyroid facing the anode end of xray machine

INTERVENTIONS:
Other: Thyroid facing the anode end of xray machine — Thyroid position: facing the anode end of xray machine
  Arms: Anode
Other: Thyroid facing the cathode end of xray machine — Thyroid position: facing the cathode end of xray machine
  Arms: Cathode

SUMMARY:
Compare the radiation in pediatric patients thyroid submitted to chest X-ray using the position of the anode and cathode.

DETAILED DESCRIPTION:
The study's primary goal was to compare radiation exposure in two different positions during chest x rays in children. It was conducted from June/2014 to July/2015, and included children from 0 to12 years old staying at the Pediatric Intensive Care Unit at the Instituto de Cardiologia de Porto Alegre, Brazil, with chest x ray requests during ICU stay. They were randomized to two groups: during the x ray, one group was positioned with the thyroid facing the anode end, and the other group was positioned with the thyroid facing the cathode end.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 12 years old
* Admitted to the Paediatric ICU at Instituto de Cardiologia de Porto Alegre
* Chest X ray requested by treating physician

Exclusion Criteria:

* Patients with scans that failed to comply with the technical criteria from the European Community Commission guidelines on quality criteria for diagnostic radiographic images in paediatrics, as evaluated by the radiologist doctors responsible for that exam report.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Dose of radiation used in thyroid gland with Ionization chamber | One month
  Assessed using ionization chamber

SECONDARY OUTCOMES:
Dose of radiation used in thorax with spectrometer | One month
  Assessed using ionization chamber
Dose of radiation used in gonads with tape to measure | One month
  Assessed using ionization chamber

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Goldmeier, Dr, Study Chair — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daruich De Souza C, Rico Freitas G, Fachel Medeiros R, Ramalho E, Rodrigues SC, Oberto Rodrigues G. Protocol for reducing radiation exposure during pediatric thoracic radiography. J Med Imaging Radiat Sci. 2022 Sep;53(3):437-443. doi: 10.1016/j.jmir.2022.05.012. Epub 2022 Jun 21. PMID 35750602
- [Derived] Rodrigues GO, Medeiros RF, Rodrigues SC, Boll LFC, Irigoyen MC, Goldmeier S. Choice of tube extremity for emission of the lowest radiation dose in pediatric patients. Int J Cardiol Heart Vasc. 2018 Oct 10;21:64-68. doi: 10.1016/j.ijcha.2018.06.006. eCollection 2018 Dec. PMID 30320204